CLINICAL TRIAL: NCT01100671
Title: Comparison of 18F-fluorodeoxyglucose Positron Emission Tomography and Coronary Computed Tomography in Assessing Vascular Inflammation in Healthy Population
Brief Title: Comparison of 18F-fluorodeoxyglucose Positron Emission Tomography and Coronary Computed Tomography in Assessing Vascular Inflammation
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Kyung Mook Choi, Professor, Korea University
Other Study IDs: PET_Coronary CT
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; vascular inflammation; MDCT; 18FDG-PET
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasam and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy patients
  Interventions: Other: Cross section study

INTERVENTIONS:
Other: Cross section study — This is not intervention study. The purpose of the study is to examine the relationship of vascular inflammation assessed by 18FDG-PET and MDCT at the cross section setting

SUMMARY:
Vascular inflammation is a key factor in both the pathogenesis and outcome of atherosclerosis. 18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) is a promising tool for identifying and quantifying vascular inflammation within atherosclerotic plaques.cardiac multidetector-row CT can provide measurements of coronary artery calcium (CAC), the degree of stenosis, and the characteristics of plaque including its potential vulnerability. Therefore, the purpose of the investigators study is to compare the usefulness of 18 FDG-PET and MDCT in assessing the vascular inflammatory status and vulnerability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients for visiting routine medical check in our clinic

Exclusion Criteria:

* History of cardiovascular disease (myocardial infarction, unstable angina, stroke, or cardiovascular revascularization)
* Diabetes
* Stage 2 hypertension (resting blood pressure, ≥ 160/100 mmHg)
* Malignancy
* Severe renal or hepatic disease
* Subjects taking medications that might affect inflammation such as NSIAD and statin

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants who underwent a medical health check in the health promotion center in Korea Guro University
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Correlation between vascular inflammatory status measured by 18FDG PET and MDCT | 20weeks

SECONDARY OUTCOMES:
Comparison the correlation with inflammatory marker and vascular inflammatory status assessed by 18FDG PET and MDCT | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mook Choi, MD.PhD, Principal Investigator — Korea University
Locations (1):
- Hye Jin Yoo, Seoul, South Korea

REFERENCES:
- [Derived] Yoo HJ, Yong HS, Hwang SY, Eo JS, Hong HC, Seo JA, Kim SG, Kim NH, Choi DS, Baik SH, Choi KM. Association of pooled cohort risk scores with vascular inflammation and coronary artery calcification in Korean adults. Metabolism. 2016 Mar;65(3):1-7. doi: 10.1016/j.metabol.2015.10.016. Epub 2015 Oct 22. PMID 26892510